CLINICAL TRIAL: NCT05950360
Title: Kinematics and Muscle Activation of Thoracic Spine and Shoulder in Rock Climbers With Shoulder Pain
Brief Title: Thoracic Spine and Shoulder Kinematics and Muscle Activation in Rock Climbers With Shoulder Pain
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Associate Professor, National Yang Ming Chiao Tung University
Other Study IDs: NYCU112095AE
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome
Keywords: Rock climbers; Shoulder pain; Shoulder impingement syndrome; Thoracic mobility; Thoracic kinematics
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome | interventions — Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- rock climbers (healthy group): Climbers without shoulder pain
  Interventions: Device: Electromagnetic tracking system, surface electromyography
- rock climbers (shoulder pain group): Climbers with shoulder pain
  Interventions: Device: Electromagnetic tracking system, surface electromyography

INTERVENTIONS:
Device: Electromagnetic tracking system, surface electromyography — arm elevation in the scapular plane, overhead reaching to the target 15° backward to the frontal plane, pull-up with overhead reaching forward and backward.

SUMMARY:
Background and Purpose: Rock climbing has been a popular sport in recent years. Rock climbing includes various open-chain and closed-chain arm movements. Overhead reaching and pull-up are the basic rock climbing elements heavily involving upper extremities. Different inclination of the wall and terrain also demand sufficient range of motion and strength of the trunk. Generally overhead reaching and arm elevation may have similar shoulder kinematics, including scapular upward rotation, posterior tilt and external rotation. Arm elevation usually is accompanied with thoracic extension and unilateral lateral flexion and rotation. During pull-up, the scapula rotates downward and externally and tilts anterior. The prevalence of shoulder injuries are about 17%, the second most common among rock climbing injuries. In the shoulder injuries, shoulder labrum lesions and shoulder impingement are the most common. Previous studies have shown that individuals with shoulder impingement syndrome have shown decreased upward and externally rotation during arm elevation, and have limited thoracic extension range of motion and greater kyphotic posture. However, a previous study found no difference in the scapular kinematics and scapular muscle activation during pull-up in rock climbers with shoulder pain and healthy climbers. The non-significant finding may be due to that the pure pull-up may not mimic climbing tasks, in which the shoulder and trunk need to adapt different inclination of the wall. Therefore, the purpose of this study is to investigate the kinematics and muscle activation of the thoracic spine and shoulder in rock climbers with shoulder pain during climbing tasks with different reaching angles. Methods: Thirty sport climbers with shoulder pain and 30 healthy climbers matched with gender, age, and dominant hand will be recruited in this study. Testing tasks will include arm elevation in the scapular plane, overhead reaching to the target 15° backward to the frontal plane, pull-up with overhead reaching forward and backward. Thoracic and shoulder kinematics will be collected using an electromagnetic tracking system. The upper trapezius, lower trapezius, serratus anterior, latissimus dorsi, and erector spinae were collected with surface electromyography (EMG). A two-way mixed ANOVA will be used to determine differences between groups in the kinematics and EMG measures at the different arm elevation angles for the testing tasks.

ELIGIBILITY:
Inclusion Criteria of Patients with Shoulder Pain:

1. Ages ranges from 18-40 years old
2. At least one year of experience of sport climbing
3. Sport Climbing frequency ≥ 6 hours per week in the last one month
4. Shoulder pain ≥ 1 month
5. Minimum of 3/10 on the numerical rating scale (NRS) in the last one month

Inclusion Criteria of Healthy Subjects in the control group:

1. Ages ranges from 18-40 years old
2. Gender, age, dominant hand and experience matching to shoulder pain climbers group
3. At least one year of experience of sport climbing
4. Sport Climbing at least 6 hours per week in the last one month
5. No history of shoulder pain in the last six months

Exclusion Criteria of Patients with Shoulder Pain and All Healthy Subjects

1. History of upper limb surgery or fracture
2. History of shoulder dislocation
3. History of neck pain, back pain, or elbow injuries in the last one year
4. Wrist or finger pain during sport climbing > 3/10 on the numerical rating scale (NRS)
5. Shoulder pain during pull-up > shoulder pain during sport climbing
6. Intensive exercise within 12 hours or any delay onset muscle soreness
7. Systemic autoimmune disease
8. Cancer
9. Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Rock climbers with and without shoulder pain
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Shoulder kinematics during arm elevation | Immediately during the experiment
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in scapular plane elevation at 30°, 60°, 90°, and 120°, and will be described with degree (°).
Thoracic kinematics during arm elevation | Immediately during the experiment
  Thoracic kinematics, including flexion, extension, side flexion and rotation in arm elevation at 30°, 60°, 90°, and 120°, and will be described with degree (°).
Shoulder kinematics during pull-up with overhead reaching forward and backward | Immediately during the experiment
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation, and will be described with degree (°).
Thoracic kinematics during pull-up with overhead reaching forward and backward | Immediately during the experiment
  Thoracic kinematics, including flexion, extension, side flexion and rotation
Scapular muscles activation during arm elevation | Immediately during the experiment
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, serratus anterior, and latissimus dorsi will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %) and calculated over three 30° increments of motion during arm elevation from 30° to 120°, including 30° - 60°, 60° - 90°, and 90° - 120°.
Trunk muscle activation during arm elevation | Immediately during the experiment
  The root mean square of electromyography (EMG) data of the erector spinae will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %) and calculated over three 30° increments of motion during arm elevation from 30° to 120°, including 30° - 60°, 60° - 90°, and 90° - 120°.
Scapular muscles activation during pull-up with overhead reaching forward and backward | Immediately during the experiment
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, serratus anterior, and latissimus dorsi will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %)
Trunk muscle activation during overhead reaching forward and backward. | Immediately during the experiment
  The root mean square of electromyography (EMG) data of the erector spinae will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %)

SECONDARY OUTCOMES:
Thoracic mobility | Immediately during the experiment
  Range of motion of thoracic spine, described with degree (°).
Thoracic kyphosis angle | Immediately during the experiment
  measured by inclinometers, described with degree (°).
Muscle length of pectoralis major | Immediately during the experiment
  In a supine position with hands behind the head. A positive (+) indicates muscle tightness, when the elbows cannot touch the testing surface.
Muscle length of pectoralis minor | Immediately during the experiment
  In a supine position, the distance between acromion and testing surface, described with cm.
Muscle length of latissimus dorsi | Immediately during the experiment
  shoulder flexion range of motion in a hook-lying position, described with degree (°)

CONTACTS AND LOCATIONS:
Overall Officials: YIN-LIANG LIN, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No